CLINICAL TRIAL: NCT06848855
Title: Evaluation of the Relationship Between Proton Pump Inhibitor Use and Dental Implant Success: a Retrospective Study
Brief Title: Proton Pump Inhibitor Use and Dental Implant Success
Status: Completed | Type: Observational
Sponsor: Berkay Tokuç (Other)
Responsible Party: Sponsor-Investigator, Berkay Tokuç, Associate Professor, Kocaeli University
Organization: Kocaeli University (Other)
Other Study IDs: 2023/295
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Implant Survival Rate; Implant Survival and Success

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the effects of proton pump inhibitors (PPIs) on the surrounding bone and the survival of dental implants. The main questions it aims to answer are:

Does PPI use affect the survival rate of dental implants? Does PPI use influence crestal bone loss and fractal dimension (FD) of the surrounding bone?

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Having a history of PPI use for more than six months,
* Having at least one bone-level and axially placed dental implant in the maxilla or mandible,
* Having a minimum of one year elapsed since the prosthetic restoration following dental implant placement,
* Having undergone routine clinical follow-ups and radiological evaluations with periapical radiographs taken using the parallel cone technique after dental implant placement.

Exclusion Criteria:

* Individuals with a history of PPI use for less than six months,
* Individuals with periapical radiographs of low image quality or with artifacts,
* Individuals for whom the regions selected for fractal analysis on periapical radiographs are not appropriately sized,
* Individuals who have not undergone routine clinical and radiographic follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted with patients who had a history of PPI use for more than six months and systemically healthy individuals who had undergone regular clinical and radiological follow-ups after dental implant placement at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Kocaeli University.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Fractal Dimension Value | Fractal analysis values were calculated on radiographs within 1 month after the data collection of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)